CLINICAL TRIAL: NCT07363200
Title: Diagnostic Agreement Between Visual Clinical Assessment and CBCT-Derived Palatal Angle Measurements for Determination of Palatal Arch Shape: Cross-Sectional Radiographic Study
Brief Title: Diagnostic Agreement Between Clinical Assessment and CBCT Palatal Angle for Palatal Arch Shape
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Adayil, Lecturer of Oral Medicine, Periodontology, and Oral Diagnosis Faculty of Dentistry, Cairo University, Cairo University
Other Study IDs: 12-25
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Morphology

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Standardized intraoral photographs corresponding to each CBCT scan will be evaluated by two calibrated examiners. Palatal arch shape will be visually classified into one of three categories: high arched palate, normal palate, or low/shallow palate. Examiners will perform assessments independently and will be blinded to CBCT measurements and to each other's results.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years
* CBCT scans showing complete hard palate
* Presence of first maxillary molars bilaterally

Exclusion Criteria:

* Palatal surgery or trauma history
* Maxillofacial anomalies
* Palatal pathology
* Poor CBCT quality

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study included adults (≥18 years) with high-quality full-maxilla CBCT scans, excluding those with craniofacial anomalies, prior palatal surgery/trauma, palatal lesions, or poor-quality images.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
diagnostic agreement of palatal shape | January 2026
  To determine the diagnostic agreement between visual clinical classification of palatal arch shape and CBCT-derived palatal angle measurements.